CLINICAL TRIAL: NCT00502008
Title: Efficacy of Coccinia Cordifolia Extract in Improving Blood Glucose Levels of Newly Diagnosed Diabetic Patients
Brief Title: Effect of Coccinia Cordifolia Extract on Blood Sugar of Newly Diagnosed Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. John's Research Institute (Other)
Collaborators: Gencor Pacific Group (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NS-2-2007
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Last update posted 2007-07-17 (Estimated); Status verified 2007-07

CONDITIONS: Diabetes
Keywords: Diabetes; India; Coccinia Cordifolia; Coccinia indica; Blood glucose levels
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Coccinia Cordifolia (herbal extract)

SUMMARY:
The purpose of the study was to evaluate the effectiveness of Coccinia Cordifolia (synonym Coccinia indica) on the blood glucose levels of newly detected type 2 diabetic patients requiring only behavioral or lifestyle intervention. The hypothesis of the study is that there will be significant decrease in the blood glucose levels after a period of 90 days in the diabetic patients who consumed the coccinia extract.

DETAILED DESCRIPTION:
The prevalence of diabetes is increasing in all countries, especially India at an alarming rate. Appropriate interventions in the form of weight reduction, changes in dietary habits and increased physical activity could help in preventing or delaying the onset of diabetes and reducing the burden due to non communicable diseases in India.

Plants or their extracts may also have a potential therapeutic role in the treatment for diabetes. Coccinia indica (synonym Coccinia cordifolia), a herb that belongs to the Cucurbitaceae family and that grows abundantly in India, is widely used in the traditional treatment of diabetes mellitus. Coccinia leaves, when administered orally twice a day for six weeks, to patients with untreated but uncomplicated maturity onset diabetes demonstrated hypoglycemic activity with significant improvement in glucose tolerance. The aim of the present study was to evaluate the effectiveness of Coccinia Cordifolia on the blood glucose levels of newly detected type 2 diabetic patients requiring only behavioral or lifestyle intervention.

The study was a double blind, placebo controlled, randomized trial. The study was carried out at Nutrition and Lifestyle Management Clinic, St. John's Medical College Hospital. After recruitment , the diabetic subjects were assigned either to the experimental or placebo group. They were provided with the extract for a period of 90 days. Prior to the intervention, the subjects underwent baseline investigations which included anthropometric, biochemical, dietary and physical activity assessment. These investigations were repeated at day 45 and day 90 of the study. The compliance of the subjects to the ingestion of capsules was documented every week when they reported to the Nutrition Clinic. All the study subjects were provided with standard dietary and physical activity advice for the control of their blood sugars. The compliance of the subjects to the prescribed diet and physical activity was assessed weekly by asking the subjects to rate their compliance on a scale of 0-100%.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinical Diagnosis of Type 2 diabetes requiring only behavioral or lifestyle intervention.
2. Fasting blood glucose in the range of 110-180 mg/dl
3. Age range - 35 to 60 years
4. Willing to participate in the study and perform all measurements

Exclusion Criteria:

1. Presence of any chronic disease or organ failure
2. Concurrent use of medication to control blood glucose levels

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2005-11; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Fasting and Post Prandial Blood Glucose, Glycosylated Hemoglobin | 90 days

SECONDARY OUTCOMES:
Serum Lipid levels | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Anura V Kurpad, MD, PhD, Principal Investigator — St. John's Research Institute
Locations (1):
- St John's Research Institute, Bangalore, Karnataka, India

REFERENCES:
- [Derived] Kuriyan R, Rajendran R, Bantwal G, Kurpad AV. Effect of supplementation of Coccinia cordifolia extract on newly detected diabetic patients. Diabetes Care. 2008 Feb;31(2):216-20. doi: 10.2337/dc07-1591. Epub 2007 Nov 13. PMID 18000183